CLINICAL TRIAL: NCT00737737
Title: Effects of Chronic Musculoskeletal Pain and Opioidergic Versus Placebo Interventions on Neuroendocrine Function in Men
Brief Title: Hormone Function in Men Treated for Pain With Opioids or Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080190; 08-NR-0190
Record Dates: First submitted 2008-08-16; First posted 2008-08-20 (Estimated); Results first posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Pain; Osteoarthritis
Keywords: Analgesia; Chronic Pain; Neuroendocrine Axis; Degenerative Diseases
MeSH Terms: conditions — Chronic Pain; Osteoarthritis; Agnosia | interventions — Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opioid (Experimental): Participants will receive MS Contin over a 4 week period starting at 15 mg bid. Doses will titrated upwards as tolerated by increments of 15-30 mg to a highest attained dose or a maximum dose of 90 mg
  Interventions: Drug: MS Contin
- Placebo (Experimental): Participants will receive a similar number of placebo tablets which match the study drug with regards to appearance over a period of 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MS Contin
  Other Names: oxycodone, morphine
  Arms: Opioid
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will examine hormone function in men with osteoarthritis pain and how it is affected by opioid medication (such as Percocet, Vicodin, MS Contin and morphine) versus placebo.

Men between 30 and 65 years of age who have had moderate to severe osteoarthritis joint pain at least 5 days a week over the past 3 months may be eligible for this study. Candidates are screened with a physical examination, x-rays, laboratory and other tests, and questionnaires about pain, mood and medical health. They are given a pain diary to complete for 2 weeks.

Participants are admitted to the hospital for two 12 hour overnight stays, during each of which they provide a 24-hour urine collection and have a small blood sample drawn every 20 minutes for 12 hours (from 8:00 p.m. to 8:00 a.m.) through a catheter that remains in place in a vein. Blood pressure and pulse are monitored during this time. After the catheter is removed, subjects complete questionnaires about their pain, mood and activity.

For the several weeks between the two hospitalizations, subjects take either an opioid medication or placebo, or standard medication such as motrin and naprosyn, according to random assignment to one of the three groups. All participants will be allowed to take anti-inflammatory medications and acetaminophen during this time as needed, but no other pain medications or treatments. They are monitored two or three times a week by telephone and complete a pain diary.

After the second hospitalization, subjects are tapered off the study medication. After 2 to 4 weeks of stopping medication, they return for a final outpatient visit to review pain or other medical problems and to have blood drawn.

DETAILED DESCRIPTION:
Use of opioid medicines for relief of chronic pain is increasing substantially but opioidergic medications and chronic pain have been both shown to perturb neuroendocrine function. The objective of this protocol is:

To determine whether long term opioid usage in men with chronic pain due to osteoarthritis results in abnormalities of Adrenocorticotropic Hormone (ACTH), cortisol, Luteinizing Hormone (LH) and testosterone secretion.

This protocol is a revised continuation of a two phase protocol with the same name which was initiated at NCCAM in 2004. In the first phase of this study 12 opioid na(SqrRoot) ve men with chronic OA pain were compared to12 healthy men by means of 12 hour overnight frequent blood sampling for measurement of baseline ACTH, cortisol, LH and testosterone. The results of phase 1 suggest that chronic osteoarthritis pain does not affect ACTH, cortisol, LH and testosterone secretion in middle aged men as compared to matched controls. In the second phase the NCCAM protocol intended to evaluate the effect of long term opioid usage AND the placebo effect if any- on the same hormones in men with chronic OA pain. Therefore the NCCAM study had a three arm design comparing MS Contin to placebo and standard treatment. When the protocol was being revised under NINR, review of the placebo literature suggested that placebo effect becomes negligible with time and therefore a two arm design was chosen comparing morphine to placebo. Baseline overnight blood hormone sampling, doses of medication, escalation and tapering schedules will be the same as in phase II of the NCCAM protocol.

Because of design changes the sample size was however recalculated to be a total of 30 opioid na(SqrRoot) ve patients with chronic OA pain. Fourteen patients, previously recruited under NCCAM, had been randomized to either morphine or placebo and finished the study. Therefore 16 additional patients need to complete the study. Taking into consideration a 25% drop out rate therefore a total of 20 patients need to be recruited. After undergoing overnight baseline hormone sampling all patients will be randomized to one of two treatment groups: MS Contin (15-90 mg), or placebo Doses of placebo and MS Contin will be escalated over 4-8 weeks in a similar fashion followed by a two-week maintenance period. At that point patients will return for repeat 12 hour frequent sampling of the same hormones as at baseline. They will then be tapered off of study medications over a period of 2-4 weeks as outpatients. Subjects will then return to clinic for a final visit and, AM blood will be obtained for ACTH, cortisol, LH, and testosterone.

The primary endpoints of this study are measures of ACTH, cortisol, LH, and testosterone secretion, whereas secondary endpoints are neurobehavioral indices such as pain symptomatology on a 0-10 (Likert) scale, the Oswestry Disability Index, Multidimensional Pain Inventory, and the Beck Depression Inventory. It is anticipated that the results of the second phase of this study will provide novel information regarding the effects of treatment with opioids on selected neuroendocrine functions in men.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Clinical evidence of chronic OA by history, examination and radiological examination

   * a. Pain level of 4/10 or greater on a scale of 0 to 10 over a 2 week screening period
   * b. Pain for a duration of 3 months or longer present at least 5 out of 7 days a week by history
   * c. Radiographic evidence of moderate to severe OA in at least one joint selected for study based on the Kellgren and Lawrence scoring scale (Appendix I:Table 2)
2. Age between 30-65 at study entry. This age range was chosen as osteoarthritis is rare in people younger than 30 and to minimize the effect of the neuroendocrine changes associated with aging on study outcome measures.
3. Men of all ethnicities
4. Ability to provide his own consent and to cooperate with study procedures
5. Willingness to refrain from drinking alcohol during the study because alcohol may exacerbate the sedative effects of morphine
6. Willingness to refrain from using muscle relaxers, antiepileptic medications and antidepressants within 6 weeks of starting study procedures
7. Willingness not to be on opioids other than prescribed by the study for the duration of the study and willingness to come off of opioids six weeks prior to starting study procedures

EXCLUSION CRITERIA:

1. Impaired pulmonary, renal, hepatic, cardiovascular or endocrine-metabolic function or major coexisting medical condition such as cancer, Cushing s disease, and diabetes which may make participation unsafe or interfere with hormone measurements
2. Prostatic disease or hypertrophy which would make subjects prone to urinary retention or require medication that would interfere with study hormone measurements
3. Sexual dysfunction including lack of libido, impotence or erectile abnormalities for safety reasons as these symptoms may be worsened by morphine
4. Rheumatoid arthritis other types of inflammatory arthritis
5. Use of systemic corticosteroids in the two months before study entry which might interfere with study hormone measurements
6. Present or past history of alcohol dependence which might predispose subjects to problems with opioid dependence based on 2 or more positive responses to the CAGE questionnaire (the latter group will be referred to psychiatry for further evaluation and excluded from study if found to fulfill psychiatric criteria for alcohol dependence or abuse)
7. Current usage of any recreational or unauthorized prescription drugs because this may indicate abuse potential based on positive urine drug test at study screening visit
8. History of opioid abuse at any time in the past based on patient report or a urine drug screen positive for opioids
9. Major depression based on a score of greater than or equal to 20 on the Beck Depression Inventory at screening, present history of major depression or treatment for major depression because these may effect endocrine function
10. Hct < 35; anemia or bleeding disorder because subjects will undergo serial blood sampling to assess hormone function
11. Allergy or inability to tolerate to morphine
12. Current or past fibromyalgia according to Wolfe criteria (1990)
13. Present or past history of sleep apnea because of increased risk of respiratory depression with morphine
14. Body mass index (BMI) > 30kg/m(2) and BMI < 20kg/m(2)
15. Local steroid injections during the study because weight has significant effects on hormone levels
16. Addition of or changes to complementary or alternative treatments during the study

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-08; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Mannes, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Joranson DE, Ryan KM, Gilson AM, Dahl JL. Trends in medical use and abuse of opioid analgesics. JAMA. 2000 Apr 5;283(13):1710-4. doi: 10.1001/jama.283.13.1710. PMID 10755497
- [Background] Bolelli G, Lafisca S, Flamigni C, Lodi S, Franceschetti F, Filicori M, Mosca R. Heroin addiction: relationship between the plasma levels of testosterone, dihydrotestosterone, androstenedione, LH, FSH, and the plasma concentration of heroin. Toxicology. 1979 Dec;15(1):19-29. doi: 10.1016/0300-483x(79)90016-7. PMID 120622
- [Background] Celani MF, Carani C, Montanini V, Baraghini GF, Zini D, Simoni M, Ferretti C, Marrama P. Further studies on the effects of heroin addiction on the hypothalamic-pituitary-gonadal function in man. Pharmacol Res Commun. 1984 Dec;16(12):1193-203. doi: 10.1016/s0031-6989(84)80084-3. PMID 6522443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with osteoarthritis at the National Institutes of Health Clinical Center. The last patient completed the study in 2012.
Pre-assignment Details: A total of 8 patients were enrolled in the study. Three patients did not qualify for the study, 1 patient elected to withdraw from the study to undergo joint surgery prior to receiving study drug and 4 patients completed the study.
Groups:
- Opioid: Participants will receive MS Contin over a 4 week period starting at 15 mg bid. Doses will titrated upwards as tolerated by increments of 15-30 mg to a highest attained dose or a maximum dose of 90 mg
  MS Contin
- Placebo: Participants will receive a similar number of matched placebo tablets over a period of 4 weeks
Period: Overall Study
Arm/Group | Opioid | Placebo
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Is Chronic Opioid Treatment Associated With Changes in Adrenocorticotropic Hormone (ACTH), Cortisol, Luteinizing Hormone (LH) and Testosterone Secretion?
Time Frame: 4 weeks
Measure: Number; unit: ng/ml
Arm/Group | Opioid | Placebo
Number analyzed (Participants) | 2 | 2
ng/ml | NA — Questionable data due to degradation of proteins to be analyzed | NA — Questionable data due to degradation of proteins to be analyzed

2. Secondary Outcome: Is Placebo Analgesia Associated With a Similar Hormonal Response as Elicited by an Opioid Analgesic?
Time Frame: 4 weeks
Measure: Number; unit: ng/ml
Arm/Group | Opioid | Placebo
Number analyzed (Participants) | 2 | 2
ng/ml | NA — Questionable data due to degradation of proteins being analyzed | NA — Questionable data due to degradation of proteins being analyzed

ADVERSE EVENTS:
Arm/Group | Opioid | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes